CLINICAL TRIAL: NCT03557190
Title: Novel Cancer Chemotherapeutics and the Vasculature: Endothelial Effects of VEGF Inhibition In Vivo in Man
Brief Title: Endothelial Effects of VEGF Inhibition In Vivo in Man
Acronym: ENDEAVOUR
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN16CA026
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases
Keywords: VEGF inhibitors; hypertension; endothelial function; thrombosis; venous occlusion plethysmography
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples without DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent developments in chemotherapy, particularly VEGF-inhibitor (VEGFI) drugs, have markedly improved the prognosis of patients with cancer. However, these drugs frequently cause high blood pressure (hypertension) which can lead to heart attacks, heart failure and stroke and can limit their use for cancer treatment.

Endothelin-1 is a hormone that causes blood vessels to tighten and may contribute to high blood pressure associated with VEGFI drugs. Blocking the effects of endothelin-1 may therefore reduce or prevent VEGFI-associated blood pressure changes, although this has never been tested in humans.

Our long-term goal is to assess the protective effects of endothelin-1 blocker drugs in patients treated with VEGFI. Before doing so, we must better explore whether VEGFIs cause blood vessel narrowing and if endothelin-1 blockers prevent this. We will assess this in healthy volunteers using a special technique called 'forearm plethysmography'. We will examine the effect of VEGFI on blood flow and also the effect of simultaneous administration of endothelin-1 blockers. These will be given at doses that produce local effects in the arm without affecting the rest of the body.

These studies study will show whether endothelin-1 blockers may help treat VEGFI-associated hypertension to enable more patients safely to receive vital cancer treatments.

DETAILED DESCRIPTION:
Developments in chemotherapy have improved the prognosis for patients with cancer.1,2 Angiogenesis is essential for tumour growth and metastasis and vascular endothelial growth factor (VEGF) is fundamental to this process.3,4 Chemotherapeutic VEGF inhibitor (VEGFI) drugs have revolutionised therapy and improved the prognosis and survival of patients with previously untreatable malignancies.1,2 Blood pressure elevation is a common complication that occurs in up to 80% of patients treated with VEGFI and almost all patients have an absolute increase in blood pressure, with 30-60% developing frank hypertension.1,5 Patients are at risk of acute hypertensive complications, including stroke, acute coronary syndrome or reversible leukoencephalopathy and the development of VEGFI-associated hypertension may mandate the premature discontinuation of these important anti-cancer therapies. Those who survive their cancer are at risk of developing end-organ damage leading to ischaemic heart disease, heart failure, renal failure and stroke.1,5 Indeed, with substantially increased cancer survivorship patients often survive long enough to allow cardiovascular morbidity to take precedence over their initial cancer diagnosis.

Mechanisms contributing to the development of VEGFI-associated hypertension may include endothelial dysfunction, capillary rarefaction and vascular remodelling.1,5 Endothelin-1 (ET-1) is a potent endogenous vasoconstrictor and is strongly implicated in the pathogenesis of hypertension and endothelial dysfunction. 3,6,7 However, the effects of VEGFI on endothelial function and the role of ET-1 in VEGFI-associated hypertension are incompletely defined. Indeed, there is a paucity of information on mechanisms contributing to VEGFI-induced hypertension and our study will address this key issue.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer male
* aged between 18 and 64 years

Exclusion Criteria:

* Unable to provide written, informed consent
* Unable or unwilling to attend for study assessments
* Current involvement in a clinical trial
* Severe or significant co-morbidity including:

  * Hypertension
  * Hyperlipidaemia
  * Cerebrovascular disease
  * Ischaemic heart disease or heart failure
  * Arial fibrillation/flutter
  * Venous or arterial thrombotic/thromboembolic event
  * Renal failure
  * Hepatic failure
* Use of any prescription medication or non-steroidal anti-inflammatory drugs within the 3 days prior to vascular assessments
* Cigarette smoker or tobacco use
* Recreational drug use
* History of anaemia
* History of cancer
* History of macular degeneration
* Ongoing inflammatory, infective or autoimmune disease
* Live vaccination received in the 3 months before the study, or expected to be required in the 6 months after the study
* Unable or unwilling to use contraception with female partners in the 6 months after the study
* BMI > 35 kg/m2
* Unable to avoid blood donation for 1 week after the study

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteer males
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow | 105 minutes
  Study drugs will be infused intra-arterially and forearm arterial blood flow assessed using forearm venous occlusion plethysmography expressed as ml per 100 ml of forearm volume per minute

SECONDARY OUTCOMES:
Change in plasma concentration of t-PA | 105 minutes
  Change in plasma concentration of t-PA measured as units/mL
Change in plasma concentration of PAI-1 | 105 minutes
  Change in plasma concentration of PAI-1 measured as units/mL

CONTACTS AND LOCATIONS:
Overall Officials: Ninian Lang, MBChB PhD, Principal Investigator — QEUH, NHS Greater Glasgow and Clyde
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided